CLINICAL TRIAL: NCT04738604
Title: Clinical Performance and Wear Resistance of Two Nano Ceramic Resin Composite in Class I Cavities: A Randomized Clinical Trial
Brief Title: Clinical Performance and Wear Resistance of Two Nano Ceramic Resin Composite in Class I Cavities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, samah mohamed bahig mohamed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91120
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Class I Dental Caries
MeSH Terms: interventions — CeramX

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany) (Active Comparator): Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany) is the ideal choice for single-tooth restorations, both in the anterior and the posterior region. It has an ultrafine, radiopaque porcelain filler for use in adhesive filling treatment. It can be polished to a high lustrer due to the ultra- fine particle filler, extremely homogeneous restorations can be placed which are easily polished to a high luster. The mechanical properties of a light-cured dental composite material are particularly dependent on its filler content, the type of incorporated fillers and the efficiency of the filler-resin coupling, so high Vickers hardness, compressive strength and flexural strength are recorded refereed to Zenit filler content 83% by weight (70% by volume) and size 0.7 microns
  Interventions: Other: Ceram•X (Dentsply De Trey GmbH, Konstanz, Germany; Other: Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany)
- Ceram•X (Dentsply De Trey GmbH, Konstanz, Germany) (Experimental): contains organically modified ceramic nanoparticles (2 to 3 nm) and nano-fillers (10 nm) that are combined with conventional glass fillers (mean particle size: 1.1 to 1.5 μm). Nanoparticles and nano-fillers comprise a polysiloxane backbone and have methacrylate groups available for polymerization. According to the manufacturer's data, filler concentration is 76% by weight and 57% by volume. Furthermore, most of the conventional resin matrix is replaced by a matrix full of highly dispersed methacrylate modified polysiloxane particles (2- 3 nm).These nano-ceramic particles are inorganic-organic hybrid particles. Both, nano-ceramic particles and nano- fillers have methacrylate groups available for polymerization. CeramX does not contain triethylene glycol dimethacrylate (TEGDMA) as it was found mutagenic and cytotoxic in vitro
  Interventions: Other: Ceram•X (Dentsply De Trey GmbH, Konstanz, Germany; Other: Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany)

INTERVENTIONS:
Other: Ceram•X (Dentsply De Trey GmbH, Konstanz, Germany — The prepared cavities will be restored with Ceram•X (Dentsply De Trey GmbH, Konstanz, Germany) with incremental placement technique (maximum: 2-mm layer). Increments will be light curing for 20 seconds according to manufacturer's instructions.
Other: Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany) — The prepared cavities will be restored with Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany) with incremental placement technique (maximum: 2-mm layer). Increments will be light curing for 40 seconds according to manufacturer's instructions.

SUMMARY:
in patients with Class I Cavities, will the use of Zenit Nano Ceramic Composite restorations have similar clinical performance to conventional Ceram-X Nano Ceramic Composite restorations, evaluation of restorations will be done at baseline, six, and twelve months using Modified USPHS Ryge criteria.

DETAILED DESCRIPTION:
The study will be conducted in the clinic of Conservative Dentistry Department, Faculty of Dentistry, Cairo University; the operator in charge samah mohamed bahig, The subjects fulfilling the eligibility criteria of the trial will be selected from the regular attendees at the clinic of Conservative Dentistry Department, Faculty of Dentistry, Cairo University. Patient examination will be done including medical history, dental history, extra-oral examination and intraoral examination. A periapical radiograph will be taken prior to restorative procedures to assess the degree of approximation of caries to pulp, intactness of lamina dura and/or presence of any periapical radiolucency to exclude the case. The field of operation will be isolated with the application of a rubber dam if possible. Otherwise, cotton rolls and the saliva ejector will be used for moisture control. For cavity preparation, local anesthetic (MepecaineL, Alexandria Company, Egypt) solution will be administrated to control patient discomfort during the procedure. The cavities will be prepared by using cylindrical #314 (Komet®, Germany) in a high speed handpiece (Sirona, Germany) rotating at high speed with copious coolant. Remaining soft caries

-if present- will be removed using sharp excavator (Maillefer, Dentsuply, Switzerland).After the cavity preparation is finished, it will be thoroughly air-water cleaned. The bonding system; the Prime and Bond universal adhesive (Dentsply De Trey GmbH, Konstanz, Germany) will be applied according to the following instructions recommended by the manufacturer and rubbed for 20 seconds then blown with a gentle air blow for 5 seconds to evaporate the solvent and then light curing for 10 seconds using LED light curing unit (>700 mW/cm2).The prepared cavities will be restored with Zenit Nano Ceramic Composite (PRESIDENT DENTAL, GmbH, Munich, Germany) will be applied with incremental placement technique (maximum: 2-mm layer). Increments will be light curing for 40 seconds according to manufacturer's instructions. and for the control group cavities will be restored withCeram•X (Dentsply De Trey GmbH, Konstanz, Germany) with incremental placement technique (maximum: 2-mm layer). Increments will be light cured for 20 seconds according to manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female gender.

  * Only co-operative patients approving to participate in the trial.
  * Good oral hygiene.
  * Medically free adult patients.
  * The age range of the patients is 20 to 54 years
  * Vital first and second molars, with Class I lesion.
  * Functioning tooth with presence of an opposing.
  * Healthy periodontium

Exclusion Criteria:

* Patients with disabilities.
* Patients having systemic diseases or severe medically compromised.
* Individuals with full dentures or crowns and bridges in occlusal contact with teeth indicated for the restorative treatment
* Pregnant or lactating subjects, or intending to become pregnant during the course of the study
* Poor oral hygiene.
* Teeth with pulpal pain.
* Teeth with periapical lesions.
* Endodontically treated teeth
* Teeth with mobility.
* Non-functioning tooth with no opposing tooth.
* Heavy occlusion or signs of severe attrition.
* Severe periodontal affection

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Anatomic form | 24 months
  Bravo: Restoration is under-contoured, without dentin or base exposure
  Charlie: Restoration is under-contoured, without dentin or base exposure.restoration need replacement.

SECONDARY OUTCOMES:
Color Match | 24 months
  Alfa: Matches tooth. Bravo: Acceptable mismatch. Charlie: Unacceptable mismatch.
Marginal Discoloration | 24 months
  Alfa: No discoloration. Bravo: minor marginal discoloration without staining toward pulp. Charlie: Deep discoloration with staining toward pulp.
Marginal Adaptation | 24 months
  Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate. Charlie: Crevice in which dentin is exposed.
Secondary Caries | 24 months
  Alfa: No active caries present. Bravo: Non-cavitated active caries is present in contact with the restoration. Charlie: Cavitated active caries is present in contact with the restoration.
Surface Texture | 24 months
  Alfa: As smooth as the surrounding enamel. Bravo: Surface rougher than enamel, clinically acceptable. Charlie: Surface unacceptably rough.
Marginal Integrity | 24 months
  Alfa: Restoration adapts closely to the tooth structure Bravo: A visible crevice. Charlie: The explorer penetrates into the crevice.
Postoperative sensitivity | 24 months
  Alfa: No post-operative sensitivity. Bravo: Short term and tolerable post-operative sensitivity. Charlie: Intolerable post-operative sensitivity.
Amount of Restoration wear. | 24 months
  Measuring unit: Microns (Quantitative)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: expecting to have all the data by October 2022

REFERENCES:
- [Derived] Bahig SM, El Sherbiney HH, Zayed MM, Ibrahim SH. A comparative 48 month randomized trial of clinical performance and wear of BISGMA based and BISGMA free nanoceramic resin composites. Sci Rep. 2025 Aug 25;15(1):31167. doi: 10.1038/s41598-025-16865-x. PMID 40850984